CLINICAL TRIAL: NCT04247269
Title: Retrospective Review of Enteral Formulas in Medically Complex Children
Brief Title: Review of Enteral Formulas in Children
Status: Withdrawn | Type: Observational
Why Stopped: Site closure due to Covid Pandemic
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 19.02.US.HCN
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2021-04

CONDITIONS: Enteral Feeding Intolerance; Tube Feeding; Nutrition Disorder, Child
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Enteral formula standard: Children fed an intact protein formula
  Interventions: Other: Enteral Tube Feeding
- Enteral formula semi-elemental: Children fed a semi-elemental protein formula
  Interventions: Other: Enteral Tube Feeding

INTERVENTIONS:
Other: Enteral Tube Feeding — Enteral tube feeding

SUMMARY:
Retrospective review of nutrition enteral formula data documented in medical records.

DETAILED DESCRIPTION:
This is a retrospective review to assess nutrition (calorie and protein) intake of enteral formula data documented in medical records of patients that consumed enteral tube feeding formulas at home.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 12 months enteral feeding
* History of enteral feeding with intact or semi-elemental formula

Exclusion Criteria:

* Medical records lacking enteral nutrition feeding use

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Population studied retrospectively will be children with a history of enteral tube feeding in a home setting and meeting inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Nutrition Intake | 12 months
  Assessment of enteral formula calorie and protein intake compared to nutrition prescription

SECONDARY OUTCOMES:
Body weight | 12 months
  Weight in kilograms
Length/height | 12 months
  Length/height (based on age) in centimeters
Formula volume consumption | 12 months
  Assessment of enteral formula volume compared to nutrition prescription
Stool frequency | 12 months
  Number of stools reported in medical record
Ventilator status | 12 months
  Assessment of ventilator change; extubated or continued

CONTACTS AND LOCATIONS:
Overall Officials: Krysmaru AraujoTorres, MD, Study Director — Société des Produits Nestlé (SPN)
Locations (1):
- Central Ohio Specialty Care, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No